CLINICAL TRIAL: NCT05000931
Title: A Pivotal, Prospective, Multi-center, Open-label Study Evaluating the Safety and Effectiveness of the CochlearTM Osia® 2 System in a Pediatric Population.
Brief Title: Osia 2 Pediatric Expansion Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: R. P. Chiacchierini Consulting, LLC (Industry); Analytical Solutions Group, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM 5766
Record Dates: First submitted 2021-07-23; First posted 2021-08-11 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Mixed Hearing Loss; Single-Sided Deafness; Conductive Hearing Loss
MeSH Terms: conditions — Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Conductive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- To demonstrate the safety of the Osia 2 System in a pediatric population aged 5 - 11 years. (Experimental)
  Interventions: Device: Osia 2 System

INTERVENTIONS:
Device: Osia 2 System — Osia 2 System in a pediatric population aged 5 - 11 years by quantifying the type, frequency and severity of adverse events.

SUMMARY:
The CochlearTM Osia®2 System was cleared by the Food and Drug Administration November 15, 2019 (K191921) for individuals aged 12 years and older who present with conductive or mixed hearing loss (up to 55 dB HL) or single-sided-deafness (SSD).Published and unpublished data suggest significant pre to postoperative benefit and minimal risk in both children and adults who have received the Osia system. Thus the objective of this study is to examine the safety and effectiveness of the Cochlear Osia 2 system in a group of pediatric subjects aged 5 to 11 years who suffer from conductive or mixed hearing loss (up to 55 dB HL), or single-sided-deafness (SSD) with the intent of expanding the indications for use.

DETAILED DESCRIPTION:
The CochlearTM Osia®2 System was cleared by the Food and Drug Administration November 15, 2019 (K191921) for individuals aged 12 years and older who present with conductive or mixed hearing loss (up to 55 dB HL) or single-sided-deafness (SSD). Published and unpublished data suggest significant pre to postoperative benefit and minimal risk in both children and adults who have received the Osia system. Due to the success of the Osia 2 system in the United States within the currently indicated patient population, clinical providers have since requested the ability to use the Osia 2 system in children aged 11 years and younger who meet the audiometric requirements. As the Osia 2 system is based on existing bone conduction and cochlear implant technologies which each possess a younger age of implantation requirement (5 years for bone conduction and 9 months for cochlear implantation), the current proposal is to align the age at implantation requirement with existing surgical bone conduction technology such as the Baha Connect and Baha Attract Systems to 5 years of age. Therefore, the objective of this study is to examine the safety and effectiveness of the Cochlear Osia 2 system in a group of pediatric subjects aged 5 to 11 years who suffer from conductive or mixed hearing loss (up to 55 dB HL), or single-sided-deafness (SSD) with the intent of expanding the indications for use.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 5 to 11 years of age with the following audiometric criterion:

   * A conductive or mixed hearing loss and still can benefit from sound amplification. The pure tone average (PTA) bone conduction (BC) threshold (measured at 0.5, 1, 2, and 3 kHz) should be better than or equal to 55 dB HL. OR
   * A profound sensorineural hearing loss in one ear and normal hearing in the opposite ear (i.e., single-sided deafness or "SSD"). The pure tone average air conduction hearing thresholds of the hearing ear should be better than or equal to 20 dB HL (measured at 0.5, 1, 2, and 3 kHz).
2. Prior experience with amplified sound through properly fitted amplification device such as a hearing aid, a CROS device, or a bone conduction device on a softband or sound arc.
3. Parent or legal guardian who is willing and able to provide written informed consent for the study participant.

Note: Subjects may include individuals seeking new implantation unilaterally (in one ear) or individuals already implanted with a bone-anchored device seeking a second-side implant (sequential bilateral)

Exclusion Criteria:

1. Insufficient bone quality or quantity to support implantation of both the BI300 Implant and the OSI200 Implant.
2. Chronic or non-revisable vestibular or balance disorders that could prevent benefit from the device, as determined by the investigator.
3. Abnormally progressive hearing loss.
4. Evidence that hearing loss is bilateral retro cochlear or bilateral central origin.
5. Evidence of conditions that would prevent speech recognition improvement as determined by the investigator.
6. Skin or scalp conditions that may preclude attachment of the Sound Processor or that may interfere with the use of the Sound Processor.
7. Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
8. Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
9. Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
10. Currently participating, or participated within the last 30 days, in another clinical investigation involving an investigational drug or device that could impact the safety or effectiveness of the Osia 2 system as determined by the investigator.
11. Individuals undergoing simultaneous single-stage aural atresia or microtia repair due to the increased risk of skin complications associated with ear reconstruction.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori O'Neill, Study Director — Cochlear
Locations (7):
- United States (7):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Children's Minnesota, Minneapolis, Minnesota
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

REFERENCES:
- [Derived] Stevens SM, Meyer A, Rivas A, Mowry S, Carvalho D, Chang KW, Germiller J, Liu YC, Tejani V. Outcomes Following Cochlear Osia 2 Implantation in Patients Ages 5-11 Years: A Multi-Center Trial. Laryngoscope. 2025 Aug;135(8):2958-2966. doi: 10.1002/lary.32159. Epub 2025 Apr 11. PMID 40214186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at seven US-based sites. The first participant was enrolled on 26 January 2022 and the last participant completed the study on 14 March 2024.
Groups:
- Implanted With the Osia 2 System: Osia 2 System in a pediatric population aged 5 - 11 years.
Period: Overall Study
Arm/Group | Implanted With the Osia 2 System
Started | 50
Completed | 49
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Implanted With the Osia 2 System
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 7 [5 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Pacific Islander | 0
  Black or African American | 2
  White | 33
  Other | 6
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Quantified by Type and Severity Between Implantation and 6-months Post-surgery.
Description: Adverse events were reported from the time of implantation through 6-months.
Time Frame: From implantation to 6 months post-surgery
Population: 1 participant withdrew after the 4-week follow-up visit.
Measure: Number; unit: Number of events
Arm/Group | Implanted With the Osia 2 System
Number analyzed (Participants) | 49
Number of events
  Adverse Device Effects | 32
  Serious Adverse Events | 8
  Serious Adverse Device Effects | 3
  Unanticipated Adverse Device Effects | 0
  Mild Events | 73
  Moderate Events | 10
  Sever Events | 4

2. Secondary Outcome: Change From Baseline to 6-months Post-surgery in SSQ (Speech, Spatial and Qualities of Hearing Scale) Parent Questionnaire
Description: Measuring change of speech, spatial, quality and conversational uses of hearing (27 items in 4 sections). Each item is scored by the parent on a scale of 0 to 10 where 0 corresponds to "not at all" and 10 to "perfectly" when rating their child's ability to hear and listen in everyday situations. The score of a participant is determined as the mean of the scores for the 4 different sections. Higher scores indicate less hearing disability.
Time Frame: Baseline before surgery, 6 months post-surgery
Population: One participant withdrew prior to the 6-month visit. One participant was unable to complete the questionnaire during the 6-month visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Implanted With the Osia 2 System
Number analyzed (Participants) | 48
score on a scale | 1.63 (1.53)

3. Secondary Outcome: Change From Baseline to 4-weeks Post-surgery in Unaided Bone Conduction Thresholds.
Description: The Pure Tone Average (PTA) is calculated as an average of the bone conduction thresholds collected at 500, 1000, 2000, and 4000 Hz. This measure was collected unaided both pre- and post-operatively to ensure no shift in bone conduction hearing as a result of the surgery.
Time Frame: Baseline before surgery, 4 weeks post-surgery
Population: 3 participants were unable to be included due to improper testing pre- and post-operatively.
Measure: Mean (Standard Deviation); unit: dB HL (decibel Hearing Level)
Arm/Group | Implanted With the Osia 2 System
Number analyzed (Participants) | 47
dB HL (decibel Hearing Level) | 0.1 (5.1)

4. Secondary Outcome: Change in Word Recognition Using Consonant Nucleus Consonant (CNC) Words Presented in Quiet From Unaided Baseline to Aided 6-months Post-surgery.
Description: The CNC Words test consists of 10 recorded lists of 50 monosyllabic words. For this study, one list is administered per test condition at 60 dBA in sound field and scored as the number of phonemes and words correct, which will be expressed as a percentage correct when analyzed. The CNC word test has a score range of 0-100% with higher values indicating better scores.
Time Frame: Baseline before surgery, 6 months post-surgery
Population: One participant withdrew prior to the 6-month visit. One participant was unable to complete the CNC word test during the baseline visit.
Measure: Mean (Standard Deviation); unit: percentage of correct words
Arm/Group | Implanted With the Osia 2 System
Number analyzed (Participants) | 48
percentage of correct words | 63.7 (24.6)

5. Secondary Outcome: Change in Sentence Recognition in Noise Using the Bramford Kowal Bench Speech-In-Noise (BKB-SIN) From Unaided Baseline to Aided 6-months Post-surgery.
Description: The Bamford-Kowal-Bench Sentence in Noise test (BKB-SIN) consists of 36 paired lists. List of sentences are presented at 65 dBA with the level of noise varied stepwise at fixed signal to noise ratio to obtain a Speech Reception Threshold (SRT) where participants are able to repeat key words 50% of the time. Score range is not specified as metric is adaptive; lower scores indicate better performance.
Time Frame: Baseline before surgery, 6 months post-surgery
Population: One participant withdrew prior to the 6-month visit. One participant was unable to complete the BKB-SIN testing during the baseline visit.
Measure: Mean (Standard Deviation); unit: db SNR (decibel Speech to Noise Ratio)
Arm/Group | Implanted With the Osia 2 System
Number analyzed (Participants) | 48
db SNR (decibel Speech to Noise Ratio) | 10.1 (7.8)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were reported from the time of implantation through 12-months post-op.
Arm/Group | Implanted With the Osia 2 System
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 7/49
Other Adverse Events (participants affected / at risk) | 23/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implanted With the Osia 2 System (N=49)
Ear Infection (Ear and labyrinth disorders) | 1
Wound dehiscence (General disorders) | 1
Tissue Breakdown (Injury, poisoning and procedural complications) | 1
Congenital Defect/Deformity (Congenital, familial and genetic disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Skin Inflammation/Irritation (Skin and subcutaneous tissue disorders) | 1
Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Implanted With the Osia 2 System (N=49)
Implant Pain (Injury, poisoning and procedural complications) | 6
Ear Infection (Ear and labyrinth disorders) | 6
Viral Infection (Infections and infestations) | 6
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 8
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has first rights to publish the multi-site data. During the study and the 12-months following the conclusion of the study, the PI may not publish or present on its own data obtained under the study. The PI may publish on their own study data (without permission from the Sponsor) or the consolidated data (with written consent from the Sponsor) by providing notice and a copy of the publication to the Sponsor at least 30 days prior to submission and allowing the Sponsor 30 days to review.

DOCUMENTS (2):
  • Study Protocol (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT05000931/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT05000931/SAP_001.pdf